CLINICAL TRIAL: NCT00998790
Title: A Post-Market Study of the AMS AdVance™ Male Sling System for the Treatment of Male Stress Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC0602
Record Dates: First submitted 2009-10-08; First posted 2009-10-20 (Estimated); Results first posted 2018-10-22 (Actual); Last update posted 2018-10-22 (Actual); Status verified 2018-01

CONDITIONS: Stress Urinary Incontinence
Keywords: Urinary Incontinence, Stress; Intrinsic sphincter deficiency; Secondary; TUR; TURP; Radical prostatectomy; Open prostatectomy; Post-suprapubic prostatectomy
MeSH Terms: conditions — Urinary Incontinence, Stress; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AMS AdVance Sling Group (Experimental): European Male subjects >40 years old who were implanted with the AMS AdVance Male Sling to treat Stress Urinary Incontinence.
  Interventions: Device: American Medical Systems (AMS) AdVance™ Male Sling System

INTERVENTIONS:
Device: American Medical Systems (AMS) AdVance™ Male Sling System — The AMS AdVance™ Male Sling System was developed to treat urinary stress incontinence in men resulting from intrinsic sphincter deficiency (ISD). The AdVance™ Male Sling System procedure is minimally invasive and consists of using two single-use needle passers and passing them through two small incisions over the obturator foramen. The needles are pushed in an arc through the tissue and exited at a perineal incision. Once the passers are through the perineal incision, the Sling System mesh arms are attached to the needles which are then pulled back through the needle track to their points of origin over the obturator foramen. The Sling System is subsequently tensioned and all incisions are closed.
  Other Names: Device: AdVance Male Sling

SUMMARY:
A prospective, multi-center study of the AdVance Male Sling for Stress Urinary Incontinence. The purpose of this study is to obtain surgical technique data for use in physician education and training and to collect early clinical outcomes data for future publication. This study is not designed to statistically demonstrate safety and efficacy of the device.

DETAILED DESCRIPTION:
A prospective, multi-center study conducted under a common implant and follow-up protocol. The study will collect pre-operative urologic testing, medical history and subject quality of life (Incontinence Quality of Life Questionaire). Intra-operative procedural data will be collected.

Pad weight and incontinence severity rating (using the ICIQ survey) will be used to characterize continence status.

Post-operative complications, urologic testing, and subject quality of life will be collected at six weeks and three, six, 12, and 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. The subject has agreed to be implanted with the AMS AdVance Male Sling System.
2. The subject is willing and able to give valid informed consent.
3. The subject is ≥40 years of age.
4. The subject has confirmed stress urinary incontinence for at least 6 months and uses no more than 8 pads per day for incontinence management and has less than 250 grams on the 24-hour pad weight test.
5. The subject has any of the following: an observable degree of incontinence during stress related activities, more than one pad is used in a 24 hour period, has more than two episodes of incontinence per day.
6. Internal sphincter contractility confirmed by endoscopic view.
7. The subject's primary etiology is TUR, TURP, or radical prostatectomy.
8. Pre-existing urological conditions, other than incontinence have been treated and are under control.
9. The subject is willing and able to return for follow-up evaluations and questionnaire completion according to the study protocol.
10. The subject is a good surgical candidate.

Exclusion Criteria:

1. The subject has a neurogenic bladder condition that is not treatable or controllable by pharmacological or alternative methods.
2. The subject has a post-void residual ≥ 100 cc.
3. The subject has detrusor-external sphincter dyssynergia.
4. The subject has a urinary tract infection (UTI).
5. The subject was treated with pelvic radiation within the last 6 months.
6. The subject currently has an inflatable penile prosthesis.
7. The subject self-catheterizes.
8. The subject has symptomatic or unstable bladder neck structure disease.
9. The subject has a history of urethral strictures that may require repetitive instrumentation.
10. The subject has previously had a urethral Sling System, an AMS Sphincter 800™, or any implanted device for the treatment of urinary incontinence (not including bulking agents).
11. The subject has a history of connective tissue or autoimmune conditions.
12. The subject has a compromised immune system.
13. The subject has renal insufficiency, and upper and/or lower urinary tract relative obstruction.
14. The subject's reading level is judged inadequate for reading and understanding the quality of life questionnaires and other study materials.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2007-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Armin Becker, MD, Principal Investigator — Oberarzt der Urologischen Klinik Grosshadern; Dirk de Ridder, Professor, Principal Investigator — UZ Gasthuisberg; Pedro Arano, MD, Principal Investigator — Fundacion Puigvert; Francois Haab, Professor, Principal Investigator — Institution Tenon Hospital; Olivier Haillot, Professor, Principal Investigator — Hopital Bretonneau; Philippe Chauveau, MD, Principal Investigator — Clinique Jules Verne; Hakim Fassi-Fehri, MD, Principal Investigator — Hopital Edouard Herriot
Locations (3):
- Universitaire Ziekenhuisen Leuven, Leuven, Belgium
- France (2):
  - Clinique Jules Verne, Nantes, Cedex 3
  - Hopital Edouard Herriot, Lyon

IPD SHARING:
Plan to Share IPD: Yes
Publications on study data currently in draft by physicians.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 114 subjects were enrolled for this study and 113 treated across 7 sites in Europe.
Period: Overall Study
Arm/Group | AMS AdVance Sling Group
Started | 114
Participants Who Were Treated | 113
Completed | 93
Not Completed | 21
Not completed — Withdrawal by Subject | 21

BASELINE CHARACTERISTICS:
Population: A total of 113 subjects were successfully implanted with the AdVance device.
Arm/Group | AMS AdVance Sling Group
Number analyzed (Participants) | 114
Age, Customized [Mean (Standard Deviation); unit: years] | 66.4 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 114
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 114
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Belgium | 31
  France | 63
  Germany | 14
  Spain | 6
Duration of Incontinence Symptoms [Mean (Standard Deviation); unit: years] | 41.8 (28.7)

OUTCOME MEASURES:

1. Primary Outcome: Change in 1-hour Pad Weight Test From Baseline to 24 Month Follow-up
Description: 1 hour pad weight tests were conducted at baseline at all successive follow-up visits. Baseline scores were compared to last visit follow-up at 24 months.
Time Frame: 24 months
Population: Baseline to 24 month measurement of 1-hour pad weight test. 113 subject available at baseline, 83 available at 24 month follow-up.
Measure: Mean (Standard Deviation); unit: grams
Groups:
- AMS AdVance Sling Group: Male subjects >40 years old who were implanted with the AMS AdVance Male Sling to treat Stress Urinary Incontinence.
Arm/Group | AMS AdVance Sling Group
Number analyzed (Participants) | 113
grams
  Baseline | 48.7 (73.4)
  24 Month Follow-up | 6.6 (17)

2. Primary Outcome: Change in 24-hour Pad Weight Test From Baseline to 24 Month Follow-up
Description: 24 hour pad weight tests were conducted at baseline at all successive follow-up visits. Baseline scores were compared to last visit follow-up at 24 months.
Time Frame: 24 months
Population: Baseline to 24 month measurement of 24-hour pad weight test. 113 subjects available at baseline, 89 available at 24 month follow-up.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | AMS AdVance Sling Group
Number analyzed (Participants) | 113
grams
  Baseline | 113.9 (79.1)
  24 Month Follow-up | 45.0 (87.6)

3. Primary Outcome: Percentage of Subjects in Each Range of Pads Per Day Use
Description: Evaluate the proportion of subjects using the following categories of pads per day from baseline to the final 24 month visit follow up 0 to 1 pads per day; 2 -3 pads per day; 4-5 pads per day; 6-7 pads per day; 8-9 pads per day; 10 or greater pads per day
Time Frame: Baseline
Measure: Number; unit: percentage of subjects
Arm/Group | AMS AdVance Sling Group
Number analyzed (Participants) | 113
percentage of subjects
  0-1 Pads Per Day | 15.9
  2-3 Pads Per Day | 66.4
  4-5 Pads Per Day | 10.6
  6-7 Pads Per Day | 6.2
  8-9 Pads Per Day | 0.9
  >10 Pads Per Day | 0

4. Primary Outcome: Percentage of Subjects in Each Range of Pads Per Day Use
Description: as for outcome 3
Time Frame: 24 months
Population: 93 subjects who completed the final 24 month follow-up visit
Measure: Number; unit: percentage of subjects
Arm/Group | AMS AdVance Sling Group
Number analyzed (Participants) | 93
percentage of subjects
  0-1 Pads Per Day | 80.6
  2-3 Pads Per Day | 12.9
  4-5 Pads Per Day | 6.5
  6-7 Pads Per Day | 0
  8-9 Pads Per Day | 0
  >10 Pads Per Day | 0

5. Secondary Outcome: To Evaluate Patient Quality of Life
Description: The Incontinence Quality of Life Questionnaire (I-QOL) is a 22 questionnaire that evaluates a subject's quality of life with respect to urinary problems/incontinence. A lower score correlates with more severe incontinence, and an increase from baseline indicates an improvement in quality of life. The score scale is 0 - 100.
  The International Consultation on Incontinence Questionnaire Short Form (ICIQ-SF) is a 4 question tool that quantifies the impact on quality of life from incontinence. A decrease from baseline to follow-up indicates an improvement in quality of life. The score scale is 0-21.
Time Frame: 24 months
Population: 113 subjects available at baseline. 90 subjects available at 24 month follow-up.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | AMS AdVance Sling Group
Number analyzed (Participants) | 113
Score on a scale
  IQOL at Baseline | 55.9 (21.6)
  IQOL at 24 Month Follow-up | 85.6 (17.3)
  ICIQ-SF at Baseline | 15.5 (3.3)
  ICIQ-SF at 24 Month Follow-up | 7.3 (5.0)

ADVERSE EVENTS:
Time Frame: All adverse events were collected during the study conductance between January 2007 through December 2012.
Description: Adverse events were collected on patients implanted with the device. One participant withdrew from the study prior to the study procedure due to not meeting inclusion/exclusion criteria.
  One hundred and twenty-three (123) adverse events in 63 subjects were reported as non-serious events. Of the 123 reported events, 70 were device related.
  Twenty-six (26) subjects experienced 36 serious adverse events; 17 of these events were device related.
Arm/Group | AMS AdVance Sling Group
Serious Adverse Events (participants affected / at risk) | 26/113
Other Adverse Events (participants affected / at risk) | 63/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AMS AdVance Sling Group (N=113)
Urinary Incontinence- Persistent (Renal and urinary disorders) | 7 (7)
Urinary Incontinence- De Novo Stres (Renal and urinary disorders) | 2 (2)
De Novo Detrusor Instability (Renal and urinary disorders) | 1 (1)
Infection- Incision Site (Renal and urinary disorders) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 1 (1)
Worsening Incontinence (Renal and urinary disorders) | 3 (3)
Hematoma (Renal and urinary disorders) | 1 (1)
Urethral Perforation (Renal and urinary disorders) | 1 (1)
Difficulty with Erections (Renal and urinary disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Other: Hernia (Musculoskeletal and connective tissue disorders) | 2 (3)
Other: Syncope/Palpitations/Heart Block (Cardiac disorders) | 2 (2)
Other: Cardiac Decompensation (Cardiac disorders) | 1 (1)
Other: Carpal Tunnel (Musculoskeletal and connective tissue disorders) | 1 (1)
Other: Chest Pain (Cardiac disorders) | 1 (1)
Other: Infection, Hernia Mesh (Infections and infestations) | 1 (1)
Other: Infection, Renal (Infections and infestations) | 1 (1)
Other: Infection, Septicemia (Infections and infestations) | 1 (1)
Other: Intestinal Hemorrhage (Gastrointestinal disorders) | 1 (1)
Other: Ischemia, Femoral (Vascular disorders) | 1 (1)
Other: Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Other: Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Other: Sub-Occlusive Syndrome, Femoral (Vascular disorders) | 1 (1)
Other: Varices (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AMS AdVance Sling Group (N=113)
Pain/Disconfort (Renal and urinary disorders) | 19 (23)
Dysuria (Renal and urinary disorders) | 8 (8)
Urinary Incontinence- De Novo Stress (Renal and urinary disorders) | 5 (5)
Urinary Incontinence- De Novo Urge (Renal and urinary disorders) | 4 (4)
Urinary Track Infection (UTI) (Renal and urinary disorders) | 7 (8)
Ecchymosis (Renal and urinary disorders) | 3 (3)
Urinary Urgency (Renal and urinary disorders) | 3 (3)
De Novo Detrusor Instability (Renal and urinary disorders) | 2 (2)
Urinary Incontinence- Persistent (Renal and urinary disorders) | 2 (2)
Urinary Retention (Renal and urinary disorders) | 2 (2)
Hematuria (Renal and urinary disorders) | 2 (2)
Post-void Dribbling (Renal and urinary disorders) | 2 (2)
Difficulty With Erections (Renal and urinary disorders) | 1 (1)
Urinary Frequency (Renal and urinary disorders) | 1 (1)
Other: Worsening Incontinence (Renal and urinary disorders) | 7 (7)
Other: Constipation (Renal and urinary disorders) | 3 (3)
Other: Catheter could not be replaced (Renal and urinary disorders) | 2 (2)
Other: Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Other: Blood Clots (Hepatobiliary disorders) | 1 (1)
Other: Coagulation at the praeputium and glans (Hepatobiliary disorders) | 1 (1)
Other: Post Void Blood Loss (Renal and urinary disorders) | 1 (1)
Other Pruritis and Swelling of Genitalia (Renal and urinary disorders) | 1 (1)
Other Scrotal Hematoma (Skin and subcutaneous tissue disorders) | 1 (1)
Other: Scrotal Numbness (Skin and subcutaneous tissue disorders) | 1 (1)
Other: Scrotal Sensitivity (Skin and subcutaneous tissue disorders) | 1 (1)
Other: Urethral Pains (Renal and urinary disorders) | 1 (1)
Other: Vein Perforation (Blood and lymphatic system disorders) | 1 (1)
Other: Influenza (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Other: Prostate Cancer (Renal and urinary disorders) | 2 (2)
Other: Syncope/Palpitations/Heart Block (Cardiac disorders) | 2 (2)
Other: Abdominal Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Other: Bacterial Infection on Penis (Renal and urinary disorders) | 1 (1)
Other: Balanitis (Renal and urinary disorders) | 1 (1)
Other: Cataract (Eye disorders) | 1 (1)
Other: Diarrhea (Gastrointestinal disorders) | 1 (1)
Other: Dry Mouth (Endocrine disorders) | 1 (1)
Other: Fatigue (General disorders) | 1 (1)
Other: Foreskin Infection (Infections and infestations) | 1 (1)
Other: Fungal Infection (Infections and infestations) | 1 (1)
Other: General Pain (General disorders) | 1 (1)
Other: Hemorrhagic Cystitis (Renal and urinary disorders) | 1 (1)
Other: Hemorrhoids (Blood and lymphatic system disorders) | 1 (1)
Other: High Blood Pressure (Cardiac disorders) | 1 (1)
Other: Inflammation of Penis (Renal and urinary disorders) | 1 (1)
Other: Itching in Pubis Area (Renal and urinary disorders) | 1 (1)
Other: Lymph Node Swelling (Endocrine disorders) | 1 (1)
Other: Nocturia (Renal and urinary disorders) | 1 (1)
Other: Parotiditis (Endocrine disorders) | 1 (1)
Other: Peripheral Edema (Vascular disorders) | 1 (1)
Other: Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Other: Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Other: Stress Incontinence (Renal and urinary disorders) | 1 (1)
Other: Stricture (Renal and urinary disorders) | 1 (1)
Other: Thyroid Lump (Endocrine disorders) | 1 (1)
Other: Ulcer (Gastrointestinal disorders) | 1 (1)
Other: Urge Incontinence (Renal and urinary disorders) | 1 (1)
Other: Wound Inflammation (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No